CLINICAL TRIAL: NCT00068861
Title: Pregnancy in Polycystic Ovary Syndrome: A 30 Week Double-Blind Randomized Trial of Clomiphene Citrate, Metformin XR, and Combined Clomiphene Citrate/Metformin XR For the Treatment of Infertility in Women With Polycystic Ovary Syndrome
Brief Title: Treatment of Infertility in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NICHD-PPCOS
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2005-09

CONDITIONS: Polycystic Ovary Syndrome; Infertility; Pregnancy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Clomiphene

INTERVENTIONS:
Drug: metformin XR
Drug: clomiphene citrate

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a common endocrine disorder affecting up to 10% of women. The primary symptoms of PCOS are menstrual irregularities, increased body and facial hair, acne, and infertility. This study will test a combination of medications in women with PCOS to determine which works best to overcome infertility.

DETAILED DESCRIPTION:
PCOS is characterized by excess circulating androgen levels and chronic anovulation. The fundamental pathophysiologic defect is unknown, but PCOS is characterized by insulin resistance and compensatory hyperinsulinemia. Improvements in insulin sensitivity in PCOS women, either through lifestyle changes or through pharmaceutical intervention, have consistently resulted in a marked improvement in the reproductive and metabolic abnormalities in PCOS. Resumption of ovulation occurs in up to 70% of women treated for PCOS. This study will evaluate the safety and effectiveness of clomiphene citrate and metformin XR in achieving a successful pregnancy in infertile PCOS women.

Women with PCOS who are seeking pregnancy will be enrolled in this study. Women will be randomized to one of three different treatment arms: A) metformin XR 1000 mg twice/day; B) clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle); or C) metformin XR 1000 mg twice/day with clomiphene citrate 50 mg/day for 5 days (day 3-7 of cycle). Women will continue on study medications for 30 weeks, 6 treatment cycles, or until they become pregnant. Progesterone levels will be drawn weekly to monitor ovulation.

ELIGIBILITY:
Inclusion Criteria

* Eight or fewer menstrual cycles in the past year or intermenstrual periods of 45 days or longer
* Elevated testosterone level
* Good general health
* Sperm concentration in partner of 20 million/ml or greater
* Ability to have intercourse 2-3 times per week
* One functional fallopian tube and normal uterine cavity

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 678
Dates: Start 2002-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Live birth rate

SECONDARY OUTCOMES:
singleton live birth rate
ovulation rate
cycles to first ovulation
cycles to conception
abortion rate
cycles to pregnancy
weeks from pregnancy to live birth

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, La Jolla, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Wayne State, Detroit, Michigan
  - University of Medicine and Dentistry New Jersey, Newark, New Jersey
  - Penn State, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Myers ER, Silva SG, Hafley G, Kunselman AR, Nestler JE, Legro RS; National Institute of Child Health and Human Development Reproductive Medicine Network. Estimating live birth rates after ovulation induction in polycystic ovary syndrome: sample size calculations for the pregnancy in polycystic ovary syndrome trial. Contemp Clin Trials. 2005 Jun;26(3):271-80. doi: 10.1016/j.cct.2005.01.006. PMID 15911461
- [Derived] Chan JL, Legro RS, Eisenberg E, Pisarska MD, Santoro N. Correlation of Polycystic Ovarian Syndrome Phenotypes With Pregnancy and Neonatal Outcomes. Obstet Gynecol. 2024 Oct 1;144(4):543-549. doi: 10.1097/AOG.0000000000005702. Epub 2024 Aug 22. PMID 39173182
- [Derived] Komorowski AS, Hughes L, Sarkar P, Aaby DA, Kumar A, Kalra B, Legro RS, Boots CE. Antimullerian hormone level predicts ovulation in women with polycystic ovary syndrome treated with clomiphene and metformin. Fertil Steril. 2024 Apr;121(4):660-668. doi: 10.1016/j.fertnstert.2023.12.031. Epub 2023 Dec 26. PMID 38154770
- [Derived] Kuang H, Jin S, Thomas T, Engmann L, Hansen KR, Coutifaris C, Casson P, Christman G, Alvero R, Santoro N, Eisenberg E, Diamond MP, Legro RS, Zhang H; Reproductive Medicine Network. Predictors of participant retention in infertility treatment trials. Fertil Steril. 2015 Nov;104(5):1236-43.e1-2. doi: 10.1016/j.fertnstert.2015.08.001. Epub 2015 Sep 3. PMID 26354094
- [Derived] Legro RS. Pregnancy in polycystic ovary syndrome I: lessons from a pragmatic explanatory with repository clinical trial. Semin Reprod Med. 2015 May;33(3):213-9. doi: 10.1055/s-0035-1552920. Epub 2015 Jun 2. PMID 26036903
- [Derived] Legro RS, Chen G, Kunselman AR, Schlaff WD, Diamond MP, Coutifaris C, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Zhang H, Foulds J; Reproductive Medicine Network. Smoking in infertile women with polycystic ovary syndrome: baseline validation of self-report and effects on phenotype. Hum Reprod. 2014 Dec;29(12):2680-6. doi: 10.1093/humrep/deu239. Epub 2014 Oct 16. PMID 25324541
- [Derived] Roth LW, Huang H, Legro RS, Diamond MP, Coutifaris C, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Zhang H, Schlaff WD; Reproductive Medicine Network. Altering hirsutism through ovulation induction in women with polycystic ovary syndrome. Obstet Gynecol. 2012 Jun;119(6):1151-6. doi: 10.1097/AOG.0b013e31825618fb. PMID 22617579
- [Derived] Aubuchon M, Kunselman AR, Schlaff WD, Diamond MP, Coutifaris C, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Legro RS; Reproductive Medicine Network. Metformin and/or clomiphene do not adversely affect liver or renal function in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Oct;96(10):E1645-9. doi: 10.1210/jc.2011-1093. Epub 2011 Aug 10. PMID 21832111
- [Derived] Schlaff WD, Zhang H, Diamond MP, Coutifaris C, Casson PR, Brzyski RG, Christman GM, Barnhart KT, Trussell JC, Krawetz SA, Snyder PJ, Ohl D, Santoro N, Eisenberg E, Huang H, Legro RS; Reproductive Medicine Network. Increasing burden of institutional review in multicenter clinical trials of infertility: the Reproductive Medicine Network experience with the Pregnancy in Polycystic Ovary Syndrome (PPCOS) I and II studies. Fertil Steril. 2011 Jul;96(1):15-8. doi: 10.1016/j.fertnstert.2011.05.069. Epub 2011 Jun 8. PMID 21645894
- [Derived] Legro RS, Schlaff WD, Diamond MP, Coutifaris C, Casson PR, Brzyski RG, Christman GM, Trussell JC, Krawetz SA, Snyder PJ, Ohl D, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Santoro N, Eisenberg E, Zhang M, Zhang H; Reproductive Medicine Network. Total testosterone assays in women with polycystic ovary syndrome: precision and correlation with hirsutism. J Clin Endocrinol Metab. 2010 Dec;95(12):5305-13. doi: 10.1210/jc.2010-1123. Epub 2010 Sep 8. PMID 20826578
- [Derived] Rausch ME, Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER, Coutifaris C; Reproductive Medicine Network. Predictors of pregnancy in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2009 Sep;94(9):3458-66. doi: 10.1210/jc.2009-0545. Epub 2009 Jun 9. PMID 19509098
- [Derived] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Ewens KG, Spielman RS, Leppert PC, Myers ER; Reproductive Medicine Network. Ovulatory response to treatment of polycystic ovary syndrome is associated with a polymorphism in the STK11 gene. J Clin Endocrinol Metab. 2008 Mar;93(3):792-800. doi: 10.1210/jc.2007-1736. Epub 2007 Nov 13. PMID 18000088
- [Derived] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER; Cooperative Multicenter Reproductive Medicine Network. Clomiphene, metformin, or both for infertility in the polycystic ovary syndrome. N Engl J Med. 2007 Feb 8;356(6):551-66. doi: 10.1056/NEJMoa063971. PMID 17287476